CLINICAL TRIAL: NCT06081270
Title: Prospective Study on Resistance-associated Mutations in Metastatic Lung Neoplasm Patients With Alterations in Driver Oncogenes, Except EGFR, Undergoing Treatment With Specific Inhibitors
Brief Title: Prospective Study on Resistance-associated Mutations in Metastatic Lung Cancer
Acronym: MUT-ONC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: MUT-ONC
Record Dates: First submitted 2023-09-06; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer
Keywords: ALK (anaplastic lymphoma kinase); ROS (ROS proto-oncogene 1); RET (Rearranged during transfection); B-RAF; lung cancer; tyrosine kinase inhibitor
MeSH Terms: conditions — Lung Neoplasms; Multiple Endocrine Neoplasia Type 2a | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Liquid biopsy — Blood withdrawal for each patient is performed (i) at the time of treatment initiation with tyrosine kinase inhibitors (TKI); (ii) at the time of the first planned instrumental re-evaluation according to clinical practice regardless of the type of response to the TKI employed (9-12 weeks); (iii) at the time of radiological progression according to RECIST 1 criteria. 1 at computerized tomography scan with contrast or metabolic progression at 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose during TKI therapy; (iv) at the time of the change of therapeutic strategy decided by the investigator when used beyond progression and not coinciding with point iii. The ctDNA is extracted from plasma and analyzed with Illumina sequencing method.

SUMMARY:
This single-centre prospective study is aimed at analysing, by means of liquid biopsy with next generation sequencing analysis on circulating tumor DNA, resistance mutations arising during therapy with selective inhibitors in patients with RTK-positive NSCLC or with mutations in the Ras/MAPK (mitogen-activated protein kinase) pathway, treated at the San Gerardo Hospital, Monza.

DETAILED DESCRIPTION:
Non-small-cell lung cancer (NSCLC) is a heterogeneous disease that may have several genetic alterations in oncogenes responsible for progression. 30-40% of NSCLC patients carry mutations affecting the Ras/MAPK pathway, while alterations in receptor tyrosine kinases (RTKs) are found in approximately 25-35% of cases. More than half of the latter are in the Epithelial Growth Factor Receptor (EGFR) gene and have been extensively studied. In the remaining cases, several genes are involved, each with lower frequencies, ranging from around 1% to 5%, depending on the studies. Despite the wide availability of inhibitors, progression remains inevitable due to the emergence of drug resistance mechanisms. The mechanisms by which resistance can be established are essentially of three types: amplification of the target gene, activation of other signal translation pathways (by-pass track) and the occurrence of mutations in the tyrosine kinase domain of the target protein. Liquid biopsy with circulating tumour DNA (ctDNA) analysis provides a non-invasive surrogate method to identify somatic mutations by means of a simple blood sample, without risk to the patient. Moreover, liquid biopsy, by collecting ctDNA from different metastatic sites, could better reflect tumour heterogeneity, both spatial and temporal, and could, therefore, constitute a simple method of longitudinal monitoring during treatment, possibly making it possible to identify relapse early before clinical manifestation. This single-centre prospective study is aimed at analysing, by means of liquid biopsy with next generation sequencing analysis on ctDNA, resistance mutations arising during therapy with selective inhibitors in patients with RTK-positive NSCLC or with mutations in the Ras/MAPK pathway, treated at the San Gerardo Hospital, Monza.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age.
2. Histological diagnosis of inoperable metastatic or locally advanced lung cancer.
3. Positivity for ALK, ROS1, MET, RET (Rearranged during transfection), NTRK (NEUROTROPHIC TYROSINE RECEPTOR KINASE) rearrangements, or KRAS (Kirsten rat sarcoma)-G12C (glycine 12 cysteine) or BRAF-V600E (valine 600 glutamate) mutations, detected by validated method (IHC Immunohistochemistry 3+, FISH (fluorescence in situ hybridization) or Next Generation Sequencing).
4. Patients undergoing radiological progression according to RECIST 1.1 criteria to treatment with generation I, II or III inhibitors in any line of treatment. Patients may also have been pre-treated with chemotherapy in earlier lines.
5. Presence of measurable disease on radiological investigations. Patients with brain metastases, even as a single site of disease, are eligible for the study.
6. Informed consent freely given and obtained before the start of the study.

Exclusion Criteria:

1. Under 18 years of age
2. Unconfirmed histological diagnosis
3. Absence of rearrangement or mutation of ALK, ROS1, MET, RET, NTRK, KRAS-G12C or BRAF-V600E
4. Progression to chemotherapy in the absence of treatment with TKI or RAS or BRAF inhibitor
5. Unmeasurable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of mutation during therapy with selective inhibitors | At treatment initiation (baseline), up to 12 weeks from treatment initiation, at the date of first documented progression, assessed up to 24 months from treatment initiation
  Evaluation of mutations in ALK (anaplastic lymphoma kinase), ROS1 (ROS proto-oncogene 1), RET, NTRK, MET, KRAS (Kirsten rat sarcoma) and BRAF and in a panel of other known oncogenes during therapy with selective inhibitors by the means of liquid biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cortinovis, MD, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori, Monza; Luca Mologni, PhD, Study Chair — University of Milano Bicocca
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared upon request
Supporting Information: CSR
Time Frame: After publication
Access Criteria: Upon request